CLINICAL TRIAL: NCT00927043
Title: Prospective, Multicenter, Epidemiological Study To Determine The Clinical, Molecular And Genetic Factors Associated To The Prognosis Of Patients With Advanced Renal Cell Carcinoma
Brief Title: Study Evaluating Renal Cell Carcinoma Risk Factors
Acronym: MICRA
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 3066K1-4433; B1771010
Record Dates: First submitted 2009-06-22; First posted 2009-06-24 (Estimated); Last update posted 2011-11-07 (Estimated); Status verified 2011-11

CONDITIONS: Carcinoma, Renal Cell
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Other: Epidemiological study according to clinical practice

INTERVENTIONS:
Other: Epidemiological study according to clinical practice — Epidemiological study according to clinical practice.

SUMMARY:
This is an epidemiological, prospective, multicenter study designed to identify the pre-treatment clinical, molecular and genetic prognostic factors associated with progression free survival in patients naïve to renal cell carcinoma (RCC) treatment.

DETAILED DESCRIPTION:
invitation to volunteer

ELIGIBILITY:
Inclusion Criteria:

* Treatment naïve patients with proven advanced RCC will be evaluated. (Except surgery or radiotherapy)
* =18 years, any gender.
* Patients with advanced Renal Cell Carcinoma and treatment naïve.

Exclusion Criteria:

* Patients who have already initiated any kind of specific therapy for the treatment of RCC.2.
* Patients with other neoplasias different from RCC (current or past).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Treatment naive patients with proven advanced RCC
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2009-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 12 months

SECONDARY OUTCOMES:
Response rate. | 12 months
Overall survival. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Pamplona, Navarre, Spain

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3066K1-4433&StudyName=Study%20Evaluating%20Renal%20Cell%20Carcinoma%20Risk%20Factors